CLINICAL TRIAL: NCT06960746
Title: Effect of Addition of Changing Lifestyle to CPAP in OSA Males Who Suffer Metabolic Syndrome and Impotence
Brief Title: Changing Lifestyle in OSA Males Who Suffer Metabolic Syndrome and Impotence: Is There a Response?
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ali Mohamed Ali ismail, lecturer of physical therapy for Cardiovascular, Respiratory disorder and Geriatrics, Faculty of Physical Therapy, Cairo University, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB00014233-31
Record Dates: First submitted 2025-04-29; First posted 2025-05-07 (Actual); Last update posted 2025-05-07 (Actual); Status verified 2025-04

CONDITIONS: Obstructive Sleep Apnea; Erectile Dysfunction; Metabolic Syndrome
MeSH Terms: conditions — Sleep Apnea, Obstructive; Erectile Dysfunction; Metabolic Syndrome

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- study group (Experimental): 20 males with metabolic syndrome, sexual impotence (erectile dysfunction), and obstructive sleep apnea will be in this group (CPAP will be applied in this group that will contain 20 males, CPAP will be applied five days weekly during night-sleeping for 4 hours for 12 weeks plus lifestyle changes that will contain 3-session per-week 40-minute treadmill exercising and low-caloric/dietary 12-week restriction.
  Interventions: Behavioral: lifestyle changing plus CPAP
- control group (Active Comparator): 20 males with metabolic syndrome, sexual impotence (erectile dysfunction), and obstructive sleep apnea will be included this control group. in this group CPAP will be applied five days weekly during night-sleeping for 4 hours for 12 weeks
  Interventions: Other: CPAP

INTERVENTIONS:
Behavioral: lifestyle changing plus CPAP — 20 males with metabolic syndrome, sexual impotence (erectile dysfunction), and obstructive sleep apnea will be in this group (CPAP will be applied in this group that will contain 20 males, CPAP will be applied five days weekly during night-sleeping for 4 hours for 12 weeks plus lifestyle changes that will contain 3-session per-week 40-minute treadmill exercising and low-caloric/dietary 12-week restriction.
  Arms: study group
Other: CPAP — 20 males with metabolic syndrome, sexual impotence (erectile dysfunction), and obstructive sleep apnea will be in this group. in this group CPAP will be applied five days weekly during night-sleeping for 4 hours for 12 weeks
  Arms: control group

SUMMARY:
The problems like metabolic syndrome and sexual impotence in males with obstructive sleep apnea are common. continuous passive airway pressure (CPAP) is an authorized treatment for this type of apnea but still the recommendations of changing lifestyles are the suggested cornerstone therapies especially in obese males

DETAILED DESCRIPTION:
Forty males with metabolic syndrome, sexual impotence (erectile dysfunction), and obstructive sleep apnea will be randomized to control group (CPAP will be applied in this group that will contain 20 males, CPAP will be applied five days weekly during night-sleeping for 4 hours for 12 weeks ) and study 20-patient group (also CPAP will be applied with the same protocol of control group plus lifestyle changes that will contain 3-session per-week 40-minute treadmill exercising and low-caloric/dietary 12-week restriction)

ELIGIBILITY:
Inclusion Criteria:

* moderate and severe obstructive sleep apnea
* erectile dysfunction (mild and moderate)
* metabolic syndrome men

Exclusion Criteria:

* cardiac patients
* psychiatric men
* autoimmune diseased men
* renal diseased men

Ages: 40 Years to 50 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — self-representation of gender identity.
Enrollment: 40 (Estimated)
Dates: Start 2025-04-15 (Actual); Primary Completion 2025-09-05 (Estimated); Study Completion 2025-09-05 (Estimated)

PRIMARY OUTCOMES:
international index of erectile function (five-item Arabic version) | it will be measured after 12 weeks
  a questionnaire that will assess erectile function

SECONDARY OUTCOMES:
index of apnea and hypopnea | It will be measured after 12 weeks
  it will assess number of events of apnea and hypapnea during one-hour sleeping
ration of oxygen desaturation per hour | It will be measured after 12 weeks
  it will assess ratio of oxygen desaturation
Epworth sleepiness scale | It will be measured after 12 weeks
  it will assess daytime sleepiness
body mass index | it will be measured after 12 weeks
  it will be measured on empty stomach
neck circumference | It will be measured after 12 weeks
  it will be measured by a tape
fasting glycemia | It will be measured after 12 weeks
  it will be assessed by blood glucose meter
high density lipoprotein | It will be measured after 12 weeks
  it will be assessed in serum
triglycerides | It will be measured after 12 weeks
  it will be assessed in serum
systolic blood pressure | It will be measured after 12 weeks
  it will be measured by manual sphygmomanometer
diastolic blood pressure | It will be measured after 12 weeks
  it will be measured by manual sphygmomanometer
waist circumference | It will be measured after 12 weeks
  it will be assessed at the level of umbilicus

CONTACTS AND LOCATIONS:
Overall Officials: Ali MA Ismail, lecturer, Principal Investigator — Cairo University
Locations (1):
- Faculty of physical therapy, Giza, Dokki, Egypt